CLINICAL TRIAL: NCT06118177
Title: Ultrasonographic Assessment of the Effects of Platelet Rich Fibrin on Wound Healing Following Palatal Connective Tissue Harvesting.
Brief Title: Ultrasonographic Assessment of Palatal Wound Healing
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gizem Torumtay Cin, assistant professor, Pamukkale University
Other Study IDs: 16.08.2022/12
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Gingival Recession; Palate; Wound
Keywords: platelet-rich fibrin; wound healing; ultrasonography; blood-flow velocity
MeSH Terms: conditions — Gingival Recession; Wounds and Injuries | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: 20-ml blood samples were taken from the antecubital vein of the patient's right or left arm in one attempt. The blood was gently transferred to glass-coated plastic tubes free from anticoagulant agents without wasting time. The tubes were immediately centrifuged at 2800 rpm for 12 min with a centrifuge device.
  After the subepithelial connective tissue graft harvesting from in the palate, obtained L-PRF was placed into donor site at the palate then incision line was suturedwith 5/0 synthetic, non-absorbable, sterile monofilament suture.
  Interventions: Procedure: connective tissue harvesting; Diagnostic Test: ultrasonography; Other: autolog platelet rich fibrin application
- Control group: After the subepithelial connective tissue graft harvesting from in the palate, the incision line was sutured with 5/0 synthetic, nonabsorbable, sterile monofilament suture. No additional material was performed into the donör area.
  Interventions: Procedure: connective tissue harvesting; Diagnostic Test: ultrasonography

INTERVENTIONS:
Procedure: connective tissue harvesting — The subepithelial connective tissue graft was obtained in each patient using the single incision technique from the region between the mesial of canine and the mesial of first molar in the palate. Connective tissue dimensions were approximately 10 × 5 × 2 mm. Finally, the incision line was sutured with 5/0 synthetic, nonabsorbable, sterile monofilament suture
Diagnostic Test: ultrasonography — A 6-18 MHz intraoral probe was used in intraoral USG examinations. Sterile gel was applied to the intraoral probe and covered with a stretch film. Then, it was placed directly on the mucosal surface of the donor site in the palatal area. Mucosal thickness was evaluated using the B-mode of the device, and vascularization was evaluated using the color doppler and pulsed wave doppler modes of the device. The following equation is used and calculated by US unit: Pulsality index (PI) = (Vmax-Vmin)/(Vmean) (Vmax is peak systolic flow velocity, Vmin is diastolic flow velocity and Vmean is mean flow velocity). The mean PI values of each patient were measured.
Other: autolog platelet rich fibrin application — Leukocyte rich PRF (L-PRF) was obtained with the centrifugation of the two tubes at 2800 rpm for 12 minutes. After centrifugation, L-PRF clots were taken from the tubes using sterile tweezers, separated from the red blood cell base using scissors. Then L-PRF membrane was placed into the donor site.
  Groups: Test group

SUMMARY:
Palatal-tissue harvesting is a routinely performed procedure in periodontal plastic surgery. Subepithelial connective tissue graft (sCTG) is considered the gold standard in root coverage. However, over the years, several materials have been attempted to accelerate wound healing and to decrease the post-operative patient discomfort and pain, which are considered the most common disadvantages of tissue harvesting from the palate. Reharvesting from the same region could be necessary in some complicated gingical recessions. For this reason, patients may face long treatment times due to recovery periods of the palate between surgeries.

Platelet-rich fibrin (PRF) which has 3-dimensional fibrin matrix structure contributes to regeneration of surgical wounds by releasing growth factors for 10-14 days and showing angiogenic properties.

In medicine and dentistry, ultrasonography (USG) method can be used to measure tissue thickness, vascularization, elasticity and blood flow. USG, as a non-invasive method, can provide objective data in evaluating the effects of surgical techniques and biomaterials used on soft tissue healing dynamics and tissue perfusion.

The investigators hypothesised that leukocyte rich PRF (L-PRF) application to the palatal area after sCTG harvesting could increase palatal tissue thickness and vascularity throughout 3-month follow-up period compared to the controls. Therefore, in this study, the investigators aimed to evaluate the effects of the L-PRF membrane on soft tissue donor site healing after harvesting sCTG in terms of wound healing dynamics using USG method.

DETAILED DESCRIPTION:
This study was planned as a randomized prospective controlled study. Patients with Miller class 1 or 2 gingival recession who needs root coverage surgery in the Department of Periodontology were included in the study. The subepithelial connective tissue graft was obtained in each patient using the single incision technique from the region between the mesial of canine and the mesial of first molar in the palate. Connective tissue dimensions were approximately 10 × 5 × 2 mm. Finally, the incision line was sutured with 5/0 synthetic, nonabsorbable, sterile monofilament suture in the control group while L-PRF membrane was placed to the donor site in the test group before the suturing. Patients were evaluated using an ultrasonography device (MyLab™ Seven, Esaote, Genoa, Italy) at the Department of Oral and Maxillofacial Radiology. USG measurements were performed on days 0, 3, 7, 14, 21, 30 and 90 for palatal tissue thickness and tissue vascularization by an oral and maxillofacial radiologist with at least six years of experience. A 6-18 MHz intraoral probe was used in intraoral USG examinations. Sterile gel was applied to the intraoral probe and covered with a stretch film. Then, it was placed directly on the mucosal surface of the donor site in the palatal area. Mucosal thickness was evaluated using the B-mode of the device, and vascularization was evaluated using the color doppler and pulsed wave doppler modes of the device. The mean pulsatility index (PI) values of each patient were calculated and considered for statistical analysis.

The power analyse of the study was performed for sample size calculation. Sample size was calculated using a statistical program (G*Power; Universitat, Dusseldorf, Germany) for α = 0.05 and effect size = 0.26. The analyses revealed that 10 subjects per group achieved a power of 80 % with 95% confidence.

The data were analysed with the SPSS 21 program (SPSS Inc., Chicago, IL). Continuous variables were presented as mean ± standard deviation and categorical variables as numbers and percentages. Shapiro-Wilk test was used to detect data's normality. For the comparison of the parameters of the study groups, independent samples T-test test was used for normally distributed data while Mann Whitney U test test was performed as non-parametric test. Within-group comparisons between the different time periods were tested with repeated measures of ANOVA. Bonferroni correction was performed for multiple variations. The statistical significance value was accepted as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Need connective tissue for tunnel operation or coronally flap operation for the treatment of gingival recession
* Non-smoking
* Good oral hygiene
* No gag reflex
* No periodontal surgery before at operation site

Exclusion Criteria:

* Systemic disorders (immunologic diseases, uncontrolled diabetes mellitus, ongoing chemotherapy or radiotherapy)
* Pregnancy/lactation/menstruation
* Inability or unwillingness to provide informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Miller 1 and 2 gingival recession who need root coverage treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
tissue thickness | at baseline before operation, on days 3, 7, 14, 21, 30, 90
  tissue thickness was measured with B-Mod mod of ultrasonography device

SECONDARY OUTCOMES:
pulsatility index | at baseline immediately after the operation, on days 3, 7, 14, 30, 90
  pulsatility index was measured with Doppler-mode of ultrasonography device

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Torumtay Cin, asist.prof., Principal Investigator — Pamukkale University Faculty of Dentistry
Locations (1):
- Pamukkale University Faculty of Dentistry, Denizli, Turkey (Türkiye)